CLINICAL TRIAL: NCT01505179
Title: The Effects of Ranolazine on Exercise Capacity in Patients With Heart Failure With Preserved Ejection Fraction
Acronym: RAZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Denise Barnard, Clinical Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN-US-259-0109; 110344 (Other: UCSD Human Research Protections Program)
Record Dates: First submitted 2011-12-08; First posted 2012-01-06 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: HFPEF; Heart Failure; HF w/ preserved EF; Preserved EF; Preserved Ejection Fraction; Diastolic Dysfunction
MeSH Terms: conditions — Heart Failure | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ranolazine (Active Comparator): Patients with be given 500 mg by mouth twice a day for three days, and then the dose will be increased to 1000 mg by mouth twice daily thereafter. (patients who concurrently take moderate CYP3A inhibitors including diltiazem, verapamil, aprepitant, erythromycin, and fluconazole will continue to 500 mg by mouth twice a day for the entire dosing period)
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Patients will be given 1 tab twice a day for 3 days, then increasing to 2 tabs twice a day thereafter (patients who concurrently take moderate CYP3A inhibitors, will be given 1 tab twice daily for the entire dosing period)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Patients with be given 500 mg by mouth twice a day for three days, and then the dose will be increased to 1000 mg by mouth twice daily thereafter. (patients who concurrently take moderate CYP3A inhibitors including diltiazem, verapamil, aprepitant, erythromycin, and fluconazole will continue to 500 mg by mouth twice a day for the entire dosing period)
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Placebo — Patients will be given 1 tab twice a day for 3 days, then increasing to 2 tabs twice a day thereafter (patients who concurrently take moderate CYP3A inhibitors, will be given 1 tab twice daily for the entire dosing period)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether treatment with Ranolazine will improve exercise capacity in patients with Heart Failure with preserved left ventricular ejection fraction, or HFPEF.

DETAILED DESCRIPTION:
Denise Barnard, M.D., and her associates, are conducting a research study to find out more about ways to improve symptoms in patients with Heart Failure with Preserved Ejection Fraction (HFPEF). Heart failure with preserved ejection fraction is a condition where the heart squeezes well but is stiff. This stiffness in the heart muscle makes the heart unable to fill, leading to shortness of breath and decreased exercise tolerance. Subjects with HFPEF are asked to participate in this study. There will be approximately 40 participants enrolled in this study. The purpose of this study is to investigate the effects of Ranolazine (Ranexa) in patients with HFPEF. The study is sponsored by the manufacturers of the drug, Gilead Pharmaceuticals.

Ranolazine is a drug that affects the ion channels in the heart. In patients with heart failure, these ion channels do not work properly, and contribute to make the heart stiff. A stiff heart leads to the symptoms of shortness of breath which patients with HFPEF experience. Due to its properties, Ranolazine may improve this stiffness. Ranolazine could improve subject's shortness of breath and ability to exercise.

Currently, ranolazine carries FDA approval for the treatment of chronic angina only. We intend to study ranolazine in patients with HFPEF, in the absence of documented ischemia, to determine whether the drug's lusitropic properties can improve exercise capacity in HFPEF patients.

Previous trials of ranolazine in patients with chronic angina found that there was a dose-dependent relationship between improvements in exercise capacity and ranolazine. However, there did appear to be a plateau in which 1500 mg of ranolazine twice daily improved exercise capacity only slightly more than 1000 mg of ranolazine given twice daily. Additionally, there was a substantially higher rate of adverse events (mainly nausea, dizziness, and asthenia) with the higher dose. Given the desire to maximize benefit and minimize the risk of adverse events, ranolazine 1000 mg by mouth twice daily was chosen as the target dose.

To properly evaluate the effects of Ranolazine, this research study is set up as a double blind, placebo controlled study. Subjects will be randomly assigned (like rolling a dice) to either Ranolazine or placebo (inactive substance). Subjects will have a 50% chance of getting the study drug and 50% chance of getting placebo.

ELIGIBILITY:
I. Inclusion Criteria

* Age > 18 years old
* Diagnosis of Heart Failure (HF) with Preserved Ejection Fraction (PEF)

  * Signs or symptoms of heart failure (breathlessness, pulmonary congestion, edema, fatigue), NYHA (New York Heart Association) Class II-III HF AND
  * LVEF (Left Ventricular Ejection Fraction) > 45% AND
  * Evidence of elevated LV filling pressures

    1. E/e-prime (E/e') mitral ratio > 8. Mitral E/e' ratio has been proposed as a noninvasive measure of left ventricular filling pressure.
    2. Brain natiuretic peptide (BNP) > 80 pg/mL. BNP is biomarker of ventricular wall stress.
* Pulmonary Artery systolic pressure estimated at > 35 mm Hg on echocardiography
* Stable medical management for at least 1 month

II. Exclusion Criteria

* Inability to perform 6 minute walk (6MW) test or 6 minute walk distance > 550 meters at baseline
* Inability to perform the Naughton protocol exercise test, or an absolute contraindication to exercise testing
* Decompensated heart failure
* Clinically significant valvular disease or congenital cardiac defects
* Clinical diagnosis of Chronic obstructive pulmonary disease (COPD) or significant lung pathology
* Prior treatment with ranolazine
* Percutaneous coronary intervention within the past 6 months or planned intervention during the study period
* Acute coronary syndrome within the prior 2 months
* Presence of uncorrected perfusion defects on stress testing
* Presence of angina
* Any rhythm other than sinus
* Electrocardiogram measured QTc interval > 500 msec
* Clinically significant hepatic impairment (ALT/AST > 3x upper limit of normal)
* Participation in another investigational drug or device study within 1 month prior to screening
* Females of childbearing potential
* Current treatment with potent inhibitors of hepatic cytochrome P450 (CYP) enzyme complex pathways affecting drug metabolism (e.g. ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, and saquinavir)
* Current treatment with CYP3A and/or P-Glycoprotein (Pgp) inducers (e.g. rifampin, rifampicin, carbamazepine, St. John's wort)
* Any other conditions that in the opinion of the investigators are likely to prevent compliance with the study protocol or pose a safety concern if the subject participates in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise D Barnard, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 12/2011 and 3/2013, the UCSD Echo database of >4500 patients (pts) and their electronic medical records were screened. Of the 1200 pts with left ventricular (LV) ejection fraction (EF) >45%, only 60 pts met all inclusion criteria. Informed consent was obtained from 10 pts who were subsequently randomized and completed study protocols.
Pre-assignment Details: Pts meeting all inclusion criteria were most often excluded due to the presence of atrial fibrillation, being unable to perform the minimum exercise effort required, or walked > 550 meters on the 6MW test. The remaining pts were excluded for acute heart failure (HF) decompensation, baseline QTc > 500 ms or participation in another clinical trial .
Groups:
- Ranolazine Group: Patients with be given 500 mg Ranolazine by mouth twice a day for three days, and then the dose will be increased to 1000 mg by mouth twice daily thereafter. (patients who concurrently take moderate CYP3A inhibitors including diltiazem, verapamil, aprepitant, erythromycin, and fluconazole will continue to 500 mg by mouth twice a day for the entire dosing period)
- Placebo Group: Patients will be given Placebo matching the appearance of Ranolazine as 1 tab twice a day for 3 days, then increasing to 2 tabs twice a day thereafter (patients who concurrently take moderate CYP3A inhibitors, will be given 1 tab twice daily for the entire dosing period)
Period: Overall Study
Arm/Group | Ranolazine Group | Placebo Group
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine Group | Placebo Group | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Full Range); unit: years] | 79.5 [63 to 82] | 75.5 [68 to 78] | 77.9 [63 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 0 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Exercise Duration [Mean (Standard Deviation); unit: seconds] — Total exercise time, measured as the duration in seconds that the subject is able to walk on a maximal effort standardized Naughton protocol treadmill test.
  seconds | 608.6 (253.1) | 328.8 (128.8) | 496.7 (206.5)
Peak Oxygen Uptake (VO2) [Mean (Standard Deviation); unit: mL O2/kg/min] — Integrative exercise performance is assessed using cardiopulmonary stress testing and expired gas analysis. The degree of reduction in peak or maximal oxygen uptake (VO2) has strong prognostic implications in HF pts. VO2 is measured as ml O2/kg/min. The modified Naughton treadmill protocol used increases the workload by approximately 3.5 ml O2/kg/min for each 2-minute stage and maximizes performance. Normally, V02 can increase from a resting value of about 3.5 ml O2/kg/min to 10-15 times the resting value.
  mL O2/kg/min | 15.9 (2.3) | 15.7 (2.1) | 15.8 (2.3)
6MW test distance [Mean (Standard Deviation); unit: meters] — The Six-minute Walk (6MW) test was designed and validated by the American Thoracic Society. It is a sub-maximal exercise test used to assess aerobic capacity and endurance. The 6MW test has the moderate ability to predict peak VO2 in patients with HF who walk less than 490 meters. Stronger correlation occurs in advanced heart failure where pts who walk less than 300 meters in 6 minutes have a low (<10 mL/kg/min) peak VO2. Normal persons average a 6MW distance of 659±62 m (range 484-820 m). Males walk on average 59±13 m further than females.
  meters | 382.5 (88.2) | 298.2 (76.3) | 348.8 (83.4)
BNP [Mean (Standard Deviation); unit: pg/mL] — Brain Natriuretic Peptide (BNP) plasma level. This biomarker reflects ventricular wall stress, often reflecting cardiac volume status or abnormal hemodynamics. Normal reference ranges are predominantly age and gender-specific but range from 0-100 pg/mL. Levels above 400 pg/ml are considered high. HF-PEF patients tend to have lower levels of BNP than patients with HF and reduced EF.
  pg/mL | 111.7 (86.4) | 184.8 (87.1) | 140.9 (86.6)
Quality of Life (QOL) Score [Mean (Standard Deviation); unit: units on a scale] — Quality of Life (QOL) in HF patients is reproducibly measured by the well-validated Minnesota Living with Heart Failure questionnaire. It is self-administered, has 21 questions and takes 5-10 minutes to complete. The test measures perceived health-related QOL. Each question is scored from 0 to 5 on the Likert scale, where 0 is 'none', and 5 is 'very much'. QOL scores range from 0 to 105; a lower score represents a better quality of life. After an intervention, a decrease in score reflects an improvement in QOL. A minimally important difference in the total score is 5 points.
  units on a scale | 36.7 (20.3) | 48.8 (36.3) | 41.5 (26.7)
Septal E/e' Doppler velocity ratio [Mean (Standard Deviation); unit: unitless] — Doppler echo allows non-invasive evaluation of diastolic cardiac function. The mitral inflow velocity (E) correlates with LV filling pressure, but is influenced by myocardial relaxation time (RT) and filling pressure. The early diastolic septal mitral annular tissue velocity (e') varies with RT alone. The unitless ratio of the E to e' velocities (E/e') is considered a reliable surrogate of LV filling pressure. Prediction of normal diastolic filling pressure is most reliable when E/e' is < 8; and of abnormal filling pressure when E/e' is > 15.
  unitless | 16.2 (3.2) | 17.0 (5.8) | 16.5 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Capacity at 6 Weeks
Description: Exercise capacity in terms of exercise duration (time in seconds) as described for the baseline value, is repeated at 6 weeks.
Time Frame: 6 weeks
Population: Entire study population
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ranolazine Group | Placebo Group
Number analyzed (Participants) | 6 | 4
seconds | 659.9 (284.5) | 300.5 (92.4)
Statistical Analysis 1: Comparison: Ranolazine Group vs Placebo Group; Test type: Superiority; p = 0.47, t-test, 2 sided

2. Primary Outcome: Change in Oxygen Consumption (VO2) at 6 Weeks
Description: Oxygen consumption (VO2) as described at baseline is remeasured after 6 weeks of drug vs placebo.
Time Frame: 6 weeks
Population: Entire study population
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Ranolazine Group | Placebo Group
Number analyzed (Participants) | 6 | 4
ml/kg/min | 17.8 (3.4) | 13.5 (4.1)
Statistical Analysis 1: Comparison: Ranolazine Group vs Placebo Group; Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Quality of Life (QOL) Score
Description: The Minnesota Living with Heart Failure (HF) Questionnaire was re-administered at the 6 week time point. The total quality of life (QOL) scores were compared to the baseline score. The well-validated Minnesota Living with Heart Failure questionnaire is self-administered, has 21 questions and takes 5-10 minutes to complete. The test measures perceived health-related QOL. Each question is scored from 0 to 5 on the Likert scale, where 0 is 'none', and 5 is 'very much'. QOL scores range from 0 to 105; a lower score represents a better quality of life. After an intervention, a decrease in score reflects an improvement in QOL. A minimally important difference in the total score is 5 points.
Time Frame: 6 weeks
Population: The analysis population is comprised of the 10 patients who were eligible and consented for participation in the trial. Six patients were assigned to the Ranolazine group and four to the placebo group, randomization was by chance.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranolazine Group | Placebo Group
Number analyzed (Participants) | 6 | 4
units on a scale | 38.2 (24.7) | 50.9 (65.5)
Statistical Analysis 1: Comparison: Ranolazine Group vs Placebo Group; Test type: Superiority; p = 0.74, t-test, 2 sided

4. Secondary Outcome: Change in Doppler Echocardiographic Parameters, Septal E/e' Ratio (E/e')
Description: Doppler echo allows non-invasive evaluation of diastolic cardiac function. The mitral inflow velocity (E) correlates with LV filling pressure, but is influenced by myocardial relaxation time (RT) and filling pressure. The early diastolic septal mitral annular tissue velocity (e') varies with RT alone. The unitless ratio of the E to e' velocities (E/e') is considered a reliable surrogate of LV filling pressure. Prediction of normal diastolic filling pressure is most reliable when E/e' is < 8; and of abnormal filling pressure when E/e' is > 15. The percent change is reported.
Time Frame: 6 weeks
Population: Entire Study Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ranolazine Group | Placebo Group
Number analyzed (Participants) | 6 | 4
percent change | -15 (35) | -1 (9.4)
Statistical Analysis 1: Comparison: Ranolazine Group vs Placebo Group; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Duration of trial, 6 weeks.
Description: The definition of adverse events and serious adverse events are not different from those found in clinicaltrials.gov definitions. The study sponsor was provided with quarterly reports regarding any/all defined AE's and SAE's for patients in our study.
  The sponsor provided us with safety letters and reports of AE/SAE's regarding ranolazine in all active clinical trials (globally).
Arm/Group | Ranolazine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 1/6 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine Group (N=6) | Placebo Group (N=4)
Minor adverse event (General disorders) | 1 (1) | 1 (1) — Headache, resolved without intervention

LIMITATIONS AND CAVEATS:
Due to slower than anticipated enrollment, only 10 subjects out of an intended 40 completed the study in the time allowed by the sponsor. The statistical analyses and inferences are restricted by low sample size and population baseline differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No